CLINICAL TRIAL: NCT04900012
Title: SPAnish DIStal PANcreatectomy Snapshot Study
Brief Title: Prospective Snapshot Audit of Distal Pancreatectomy in Spain
Acronym: Spadispan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Candido Fernando Alcazar-Lopez, MD PHD Senior consultant HPB surgeon, Hospital General Universitario de Alicante
Other Study IDs: 2021/078
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Surgery--Complications; Pancreas Disease; Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Distal pancreatectomy: All cases operated on performing distal pancreatectomy in involved Units
  Interventions: Procedure: Distal pancreatectomy

INTERVENTIONS:
Procedure: Distal pancreatectomy — We are going to collect all cases
  Other Names: corporocaudal pancreatectomy

SUMMARY:
Distal pancreatectomy is the surgical technique performed to treat many pancreatic diseases located in neck and tail of the pancreas. Laparoscopic approach is the gold standard but in many centres the percentage of laparoscopic approach is still low. This technique has low mortality but 30% morbidity mostly related to pancreatic fistula. Some new devices (linear stapler, energy devices and patches) seem to decrease pancreatic fistula but there is not evidence based medicine that confirm the results published usually in unicentric studies.

DETAILED DESCRIPTION:
Snapshot observational study including most of the Spanish pancreatic units that perform distal pancreatectomy. One year consecutive cases.

Main objectives.

1. percentage of laparoscopic approach in Spain
2. Morbidity at 90 days measured by CCI and Clavien Dindo
3. Percentage of pancreatic fistula
4. Impact of new device to decrease pancreatic fistula

ELIGIBILITY:
Inclusion Criteria:

-All distal pancreatectomies performed in involved Units

Exclusion Criteria:

* No sign of informed consent for entering in the study
* Emergency procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All scheduled distal pancreatectomies performed in on year in each Unit.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity at 90 days | 90 days
  Morbidity measured with CCI and Clavien at 90 days
Laparoscopic approach | 1 year
  Laparoscopic or laparotomy approach

SECONDARY OUTCOMES:
Pancreatic fistula | 90 days
  Percentage of pancreatic fistula

IPD SHARING:
Plan to Share IPD: No
CRD is done. It should be sent to local investigators and fulfilled in a Castor formulary.